CLINICAL TRIAL: NCT04524351
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of Posiphen® in Subjects With Early Alzheimer's Disease (AD) or Early Parkinson's Disease (PD)
Brief Title: Posiphen® Dose-Finding, Biomarker Study in Early Alzheimer's and Parkinson's Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Annovis Bio Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANVS-12003
Record Dates: First submitted 2020-08-11; First posted 2020-08-24 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease; Parkinson Disease
Keywords: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Neurotoxic proteins; Neurotransmitters; Amyloid Precursor Proteins; Inflammatory factors; Synaptic factors; CSF
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease | interventions — phenserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Posiphen, 80mg (Parkinson's Participants) (Active Comparator): Posiphen Oral Capsule, 80mg, taken once per day for 25±2 days.
  Interventions: Drug: Posiphen
- Posiphen, 40mg (Parkinson's Participants) (Active Comparator): Posiphen Oral Capsule, 40mg, taken once per day for 25±2 days.
  Interventions: Drug: Posiphen
- Posiphen, 20mg (Parkinson's Participants) (Active Comparator): Posiphen Oral Capsule, 20mg, taken once per day for 25±2 days.
  Interventions: Drug: Posiphen
- Posiphen, 10mg (Parkinson's Participants) (Active Comparator): Posiphen Oral Capsule, 10mg, taken once per day for 25±2 days.
  Interventions: Drug: Posiphen
- Posiphen, 5mg (Parkinson's Participants) (Active Comparator): Posiphen Oral Capsule, 5mg, taken once per day for 25±2 days.
  Interventions: Drug: Posiphen
- Placebo (Parkinson's Participants) (Placebo Comparator): Placebo Oral Capsule, taken once per day for 25±2 days.
  Interventions: Drug: Placebo
- Placebo (Alzheimer's Participants) (Placebo Comparator): Placebo Oral Capsule, taken once per day for 25±2 days.
  Interventions: Drug: Placebo
- Posiphen, 80mg (Alzheimer's Participants) (Active Comparator): Posiphen Oral Capsule, 80mg, taken once per day for 25±2 days.
  Interventions: Drug: Posiphen

INTERVENTIONS:
Drug: Posiphen — Solid oral dosage form, capsule
  Arms: Posiphen, 10mg (Parkinson's Participants); Posiphen, 20mg (Parkinson's Participants); Posiphen, 40mg (Parkinson's Participants); Posiphen, 5mg (Parkinson's Participants); Posiphen, 80mg (Alzheimer's Participants); Posiphen, 80mg (Parkinson's Participants)
Drug: Placebo — Solid oral dosage form, capsule
  Arms: Placebo (Alzheimer's Participants); Placebo (Parkinson's Participants)

SUMMARY:
Annovis is conducting a clinical study to investigate Posiphen in patients with Early Alzheimer's Disease (AD) and Early Parkinson's Disease (PD). Investigators are looking to recruit 68 patients in two parts of the study. In Part one of the study Investigators will recruit 14 AD and 14 PD patients who will either receive placebo (an inert pill which looks like the study drug) or the study drug Posiphen, both taken daily. In Part two of the study Investigators will recruit 40 PD patients who will receive different strengths of the study drug Posiphen taken daily. Patients will be required to come to the site for 3 face to face visits and have 4 phone calls, tests include but are not limited to, blood and CSF (spinal fluid) sampling, cognitive assessments, clinical examinations and laboratory safety tests. Primarily the Investigators are looking for the safety and tolerability of Posiphen, although Investigators will also evaluate the activity of Posiphen by a number of different biomarkers measuring pathway and target engagements.

DETAILED DESCRIPTION:
Part 1 is a study with 14 Early AD and 14 Early PD patients who are randomized to 80 mg of Posiphen or placebo. Participants will undergo a Screening Visit, provide informed consent and be evaluated for eligibility per the inclusion and exclusion criteria. If enrolled, participants will proceed to the randomized treatment portions of the study. Period 1 consists of first-time dosing in clinic with administration of 80 mg of Posiphen or Placebo. Period 2 consists of an at home dosing period of 25±2 days, with daily administration of 80 mg of Posiphen or Placebo. Period 3 will be comprised of a stay at the clinical research unit where the subject will undergo study procedures that include safety assessments (AE and concomitant medication monitoring, 12-lead ECGs, clinical laboratory testing, vital signs assessments, and physical examinations), the last dose of Posiphen or Placebo, and 6 hours of blood and CSF sampling. At the end of blood/CSF sampling, the subjects will need to stay for a minimum of 1 hour of observation but may stay if necessary for observation until the following day (e.g., if the subject has blood/CSF sampling on Day 25, he/she may stay for observation until Day 26). After all end-of-study procedures are complete, the subject will be discharged to home. A 24-hour follow-up call will occur to assess the participants current condition and if there are any additional adverse events to report.

After completion of Part 1 of the study, the plasma and CSF samples will be analyzed for the biomarkers to determine if changes are needed to the biomarkers to be measured in Part 2. Since the conduct of the study in Part 2 will be identical to the conduct of the study in Part 1, recruitment will continue uninterrupted. The only potential change between Part 1 and Part 2 are the biomarkers to be measured.

Part 2 is a study with 40 Early PD patients, 10 patients each who are randomized to one of 4 treatment conditions of Posiphen (5 mg, 10 mg, 20 mg, or 40 mg). Participants will undergo a Screening Visit, provide informed consent and be evaluated for eligibility per the inclusion and exclusion criteria. If enrolled, participants will proceed to the randomized treatment portions of the study. Period 1 consists of first-time dosing in clinic with administration of 5, 10, 20, or 40mg of Posiphen. Period 2 consists of an at home dosing period of 25±2 days, with daily administration of 5, 10, 20, or 40mg of Posiphen. Period 3 will be comprised of a stay at the clinical research unit where the subject will undergo study procedures that include safety assessments (AE and concomitant medication monitoring, 12-lead ECGs, clinical laboratory testing, vital signs assessments, and physical examinations), the last dose of Posiphen or Placebo, and 6 hours of blood and CSF sampling. At the end of blood/CSF sampling, the subject will need to stay for a minimum of 1 hour of observation but may stay if necessary for observation until the following day (e.g., if the subject has blood/CSF sampling on Day 25, he/she may stay for observation until Day 26). After all end-of-study procedures are complete, the subject will be discharged to home. A 24-hour follow-up call will occur to assess the participant's current condition and if there are any additional adverse events to report.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet the following criteria:

1. Male or female aged 45 years and over.
2. Female participants must be of non-childbearing potential or post-menopausal for at least 2 consecutive years or surgically sterile (bilateral tubal ligation, hysterectomy or bilateral oophorectomy) for at least 6 months prior to screening.
3. Female participants will be given a urine pregnancy test at the screening visit for which they should test negative.
4. A) AD - CDR = 0.5 or 1. B) PD - Hoehn & Yahr ≤ 4; PD criteria by MDS-UPDRS.
5. A) AD MMSE score between the range of 18 to 28. B) PD MMSE score between the range of 18 to 30.
6. General cognition and functional performance sufficiently preserved that the subject can provide written informed consent.
7. No evidence of current suicidal ideation or previous suicide attempt in the past month as evaluated in the Columbia Suicide Severity Rating Scale.
8. MRI scan within the 12 months prior to screening without evidence of infection, infarction, or other focal lesions and without clinical symptoms suggestive of intervening neurological disease. Lacunes that are not believed to contribute to the subject's cognitive impairment are permissible. If there is no MRI available within a 12-month timeframe, then an MRI must be performed as part of the screening procedures for eligibility.
9. Stability of permitted medications prior to screening.

   1. Stable for at least 12 weeks: Cholinesterase inhibitors and/or memantine medication
   2. Stable for at least 4 weeks:

   i. Anti-parkinsonian medication ii. Anticonvulsant medications used for epilepsy or mood stabilization; neuropathic pain indications iii. Mood-stabilizing psychotropic agents, including, but not limited to, lithium.
10. Adequate visual and hearing ability (physical ability to perform all the study assessments).
11. Good general health with no disease expected to interfere with the study.
12. Subjects previously exposed to Posiphen may be included in the study.

Exclusion Criteria

Subjects meeting any of the following criteria must not be included in the study:

1. Has a history of a psychiatric disorder such as schizophrenia, bipolar disorder or major depression according to the criteria of the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM). Mild depression or history of depression that is stable on treatment with a SSRI or SNRI medication at a stable dose is acceptable.
2. History of a seizure disorder.
3. Has a history or current evidence of long QT syndrome, Fridericia's formula corrected QT (QTcF) interval ≥ 450ms, or torsades de pointes.
4. Has bradycardia (<50 bpm) or tachycardia (>100 bpm) on the ECG at screening.
5. Has uncontrolled Type-1 or Type-2 diabetes . A Subject with HbA1c levels up to 7.5% can be enrolled if the investigator believes the subject's diabetes is under control.
6. Has clinically significant renal or hepatic impairment.
7. Has any clinically significant abnormal laboratory values. Subjects with liver function tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) greater than twice the upper limit of normal will be excluded.
8. Is at imminent risk of self-harm, based on clinical interview and responses on the C SSRS, or of harm to others in the opinion of the Investigators. Subjects must be excluded if they report suicidal ideation with intent, with or without a plan or method (e.g. positive response to Items 4 or 5 in assessment of suicidal ideation on the C SSRS) in the past 2 months, or suicidal behavior in the past 6 months.
9. Has four or more signal hypointensities on T2*-weighted gradient recalled echo magnetic resonance sequences that are thought to represent hemosiderin deposits including microhemorrhages and superficial siderosis or evidence of acute or sub-acute micro or microhemorrhage as noted on the MRI scan.
10. Has cancer or has had a malignant tumor within the past year, except patients who underwent potentially curative therapy with no evidence of recurrence. (Patients with stable untreated prostate cancer or skin cancers are not excluded).
11. Alcohol / Substance use disorder, moderate to severe, in the last 5 years according to the most current version DSM.
12. Participation in another clinical trial with an investigational agent and have taken at least one dose of study medication, unless unblinded on placebo, within 60 days prior to the start of screening. (The end of a previous investigational trial is the date the last dose of an investigational agent was taken), or five half-lives of the investigational drug, whichever is greater.
13. Subjects with infection or inflammation of the skin or skin disease at or in proximity to the lumbar puncture site.
14. History of lumbar spine surgery or chronic low back pain (CLBP).
15. Subjects with learning disability or developmental delay.
16. Subjects whom the site PI deems to be otherwise ineligible.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - New England Institute for Clinical Research, Stamford, Connecticut
  - DeLand Clinical Research Unit, DeLand, Florida
  - MD Clinical, Hallandale, Florida
  - Homestead Associates in Research, Miami, Florida
  - Ezy Medical Research Co., Miami, Florida
  - Conquest Research LLC, Winter Park, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Quest Research Institute, Farmington Hills, Michigan
  - North Suffolk Neurology, PC, Port Jefferson Station, New York
  - Penn Medicine, Department of Neurology, U of PA, Philadelphia, Pennsylvania
  - University of Texas Health Science Center, San Antonio, Texas
  - Aspen Clinical Research LLC, Orem, Utah

REFERENCES:
- [Derived] Fang C, Hernandez P, Liow K, Damiano E, Zetterberg H, Blennow K, Feng D, Chen M, Maccecchini M. Buntanetap, a Novel Translational Inhibitor of Multiple Neurotoxic Proteins, Proves to Be Safe and Promising in Both Alzheimer's and Parkinson's Patients. J Prev Alzheimers Dis. 2023;10(1):25-33. doi: 10.14283/jpad.2022.84. PMID 36641607

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posiphen, 80mg (Parkinson's Participants) | Posiphen, 40mg (Parkinson's Participants) | Posiphen, 20mg (Parkinson's Participants) | Posiphen, 10mg (Parkinson's Participants) | Posiphen, 5mg (Parkinson's Participants) | Placebo (Parkinson's Participants) | Placebo (Alzheimer's Participants) | Posiphen, 80mg (Alzheimer's Participants)
Started | 10 | 10 | 11 | 10 | 12 | 5 | 6 | 10
Completed | 9 | 9 | 11 | 9 | 11 | 5 | 5 | 10
Not Completed | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posiphen, 80mg (Parkinson's Participants) | Posiphen, 40mg (Parkinson's Participants) | Posiphen, 20mg (Parkinson's Participants) | Posiphen, 10mg (Parkinson's Participants) | Posiphen, 5mg (Parkinson's Participants) | Placebo (Parkinson's Participants) | Placebo (Alzheimer's Participants) | Posiphen, 80mg (Alzheimer's Participants) | Total
Number analyzed (Participants) | 10 | 10 | 11 | 10 | 12 | 5 | 6 | 10 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (9.31) | 62.5 (6.74) | 69.8 (10.93) | 62.0 (9.93) | 67.2 (6.94) | 75.4 (3.13) | 68.0 (6.87) | 72.8 (6.34) | 67.3 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 3 | 2 | 2 | 3 | 8 | 25
  Male | 8 | 8 | 8 | 7 | 10 | 3 | 3 | 2 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 5 | 2 | 3 | 2 | 4 | 5 | 21
  Not Hispanic or Latino | 10 | 10 | 6 | 8 | 9 | 3 | 2 | 5 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  White | 10 | 10 | 9 | 10 | 12 | 5 | 4 | 8 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 11 | 10 | 12 | 5 | 6 | 10 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events
Description: Percent of patients with AEs in the Posiphen treatment arms compared to the Placebo group
Time Frame: 25±2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Posiphen, 80mg (Parkinson's Participants) | Posiphen, 40mg (Parkinson's Participants) | Posiphen, 20mg (Parkinson's Participants) | Posiphen, 10mg (Parkinson's Participants) | Posiphen, 5mg (Parkinson's Participants) | Placebo (Parkinson's Participants) | Placebo (Alzheimer's Participants) | Posiphen, 80mg (Alzheimer's Participants)
Number analyzed (Participants) | 10 | 10 | 11 | 10 | 12 | 5 | 6 | 10
Participants | 3 | 5 | 4 | 6 | 1 | 3 | 3 | 5

2. Secondary Outcome: Concentration of Posiphen in Plasma
Description: Maximum Plasma Concentration (Cmax) of Posiphen reported as ng/mL.
Time Frame: Samples collected over a 6 hour timeframe
Population: Samples successfully collected for PK measurement were analyzed. Some participants did not provide sufficient samples for analysis. Placebo participants were not analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posiphen, 80mg (Parkinson's Participants) | Posiphen, 40mg (Parkinson's Participants) | Posiphen, 20mg (Parkinson's Participants) | Posiphen, 10mg (Parkinson's Participants) | Posiphen, 5mg (Parkinson's Participants) | Placebo (Parkinson's Participants) | Placebo (Alzheimer's Participants) | Posiphen, 80mg (Alzheimer's Participants)
Number analyzed (Participants) | 9 | 9 | 11 | 9 | 8 | 0 | 0 | 9
ng/mL | 94.9 (33.4) | 40.2 (19.7) | 15.3 (21.6) | 2.0 (1.4) | 0.4 (0.3) |  |  | 112.3 (49.3)

3. Other Pre Specified Outcome: Change in Abeta42/Abeta40 Ratio
Description: Biomarker related to neurotoxic protein cascade measured in patient sample
Time Frame: Baseline to 25±2 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Changes in Functional Impairment
Description: Functional impairment will be evaluated using the Clinical Dementia Rating (CDR) scale (Berg1988) for AD.
Time Frame: Baseline to 25±2 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes in Functional Impairment
Description: Functional impairment will be evaluated using the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) scale (Goetz 2008) for those with PD.
Time Frame: Baseline to 25±2 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Cognition
Description: For both populations, the Mini-Mental State Examination (MMSE) scale (Folstein 1975) will be administered as a global measure of cognition.
Time Frame: Baseline to 25±2 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Cognition
Description: For both populations, the Coding subtest from the Weschler Adult Intelligence Scales, 4th edition (WAIS-IV) will serve as a sensitive measure of CNS dysfunction.
Time Frame: Baseline to 25±2 days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Cognition
Description: The subjects with AD will also be administered the The Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) Subscale (Schafer 2012).
Time Frame: Baseline to 25±2 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 25±2 days
Arm/Group | Posiphen, 80mg (Parkinson's Participants) | Posiphen, 40mg (Parkinson's Participants) | Posiphen, 20mg (Parkinson's Participants) | Posiphen, 10mg (Parkinson's Participants) | Posiphen, 5mg (Parkinson's Participants) | Placebo (Parkinson's Participants) | Placebo (Alzheimer's Participants) | Posiphen, 80mg (Alzheimer's Participants)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/10 | 0/12 | 0/5 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/10 | 0/12 | 0/5 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 5/10 | 4/11 | 6/10 | 1/12 | 3/5 | 3/6 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posiphen, 80mg (Parkinson's Participants) (N=10) | Posiphen, 40mg (Parkinson's Participants) (N=10) | Posiphen, 20mg (Parkinson's Participants) (N=11) | Posiphen, 10mg (Parkinson's Participants) (N=10) | Posiphen, 5mg (Parkinson's Participants) (N=12) | Placebo (Parkinson's Participants) (N=5) | Placebo (Alzheimer's Participants) (N=6) | Posiphen, 80mg (Alzheimer's Participants) (N=10)
puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
electrocardiogram QT prolongation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1
headache (Nervous system disorders) | 0 | 1 | 3 | 4 | 0 | 1 | 0 | 2
cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
movement disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
fatigue (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
catheter site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
procedural headache (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
uppper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
urine analysis abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT04524351/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT04524351/SAP_002.pdf